CLINICAL TRIAL: NCT03261427
Title: A Randomized, Open-label, Phase I Clinical Trial to Evaluate the Pharmacokinetic Characteristics and Safety/Tolerability of YNP-1807 Compared to Lyrica® After Oral Administration in Healthy Adult Volunteers: Part I- Single Dosing/Part II- Multiple Dosing
Brief Title: Evaluate the Pharmacokinetic Characteristics and Safety/Tolerability of YNP-1807 Compared to Lyrica® After Oral Administration Adult Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yungjin Pharm. Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: YJ16-101
Record Dates: First submitted 2017-08-22; First posted 2017-08-25 (Actual); Last update posted 2019-07-10 (Actual); Status verified 2019-07

CONDITIONS: Healthy
MeSH Terms: interventions — Pregabalin; Tablets

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- YNP-1807 Tablet(Pregabalin 330mg) (Experimental): YNP-1807(Pregabalin 330mg), QD
  Interventions: Drug: YNP-1807 330Mg Tablet
- Lyrica Capsule(Pregabalin 150mg) (Active Comparator): Lyrica Capsule(Pregabalin 150mg), BID
  Interventions: Drug: Lyrica 150Mg Capsule

INTERVENTIONS:
Drug: Lyrica 150Mg Capsule — 150 mg oral administered (BID)
  Arms: Lyrica Capsule(Pregabalin 150mg)
Drug: YNP-1807 330Mg Tablet — 330 mg oral administered (QD)
  Arms: YNP-1807 Tablet(Pregabalin 330mg)

SUMMARY:
The purpose of this trial to compare the pharmacokinetic characteristics of YNP-1807(Pregabalin 330mg) and Lyrica capsule(Pregabalin 150mg). YNP-1807 is made by Yungjin Pharm. Primary endpoints are AUClast and Cmax and secondary endpoints are AUCinf, Tmax, t1/2, Vd/f, CL/f.

ELIGIBILITY:
Inclusion Criteria:

* 19 years to 55 years healthy volunteers adult at screening visit
* For male, weight is more than 55 kg, for female, weight is more than 50 kg.
* Body mass index(BMI) value : 18.5 to 25.0 kg/m2
* If female, should be included one at least as following

  * menopausal(menstruation for 2 years minimum)
  * surgery infertility

Exclusion Criteria:

* Any history of drug overdose or dependence
* Female who is pregnant or nursing
* AST, ALT > ULN*1.25
* Total bilirubin > ULN*1.5
* CPK > ULN*1.5

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2017-09-14 (Actual); Primary Completion 2017-10-11 (Actual); Study Completion 2018-03-29 (Actual)

PRIMARY OUTCOMES:
Part I : AUClast of Pregabalin | 0,1,2,3,4,5,6,7,8,10,12,16,20,24,36 hours
Part I : Cmax of Pregabalin | 0,1,2,3,4,5,6,7,8,10,12,16,20,24,36 hours
Part II : AUCτ,ss of Pregabalin | Pre-dose, 0,1,2,3,4,5,6,7,8,10,12,16,20,24,36 hours
Part II : Cmax,ss of Pregabalin | Pre-dose, 0,1,2,3,4,5,6,7,8,10,12,16,20,24,36 hours

SECONDARY OUTCOMES:
Part I : AUCinf of Pregabalin | 0,1,2,3,4,5,6,7,8,10,12,16,20,24,36 hours
Part I : Tmax of Pregabalin | 0,1,2,3,4,5,6,7,8,10,12,16,20,24,36 hours
Part I : t1/2 of Pregabalin | 0,1,2,3,4,5,6,7,8,10,12,16,20,24,36 hours
Part I : Vd/F of Pregabalin | 0,1,2,3,4,5,6,7,8,10,12,16,20,24,36 hours
Part I : CL/F of Pregabalin | 0,1,2,3,4,5,6,7,8,10,12,16,20,24,36 hours
Part II : Cmin,ss of Pregabalin | Pre-dose, 0,1,2,3,4,5,6,7,8,10,12,16,20,24,36 hours
Part II : AUClast,ss of Pregabalin | Pre-dose, 0,1,2,3,4,5,6,7,8,10,12,16,20,24,36 hours
Part II : Tmax,ss of Pregabalin | Pre-dose, 0,1,2,3,4,5,6,7,8,10,12,16,20,24,36 hours
Part II : t1/2 of Pregabalin | Pre-dose, 0,1,2,3,4,5,6,7,8,10,12,16,20,24,36 hours
Part II : CLss/F of Pregabalin | Pre-dose, 0,1,2,3,4,5,6,7,8,10,12,16,20,24,36 hours
Part II : Vdss/F of Pregabalin | Pre-dose, 0,1,2,3,4,5,6,7,8,10,12,16,20,24,36 hours
Part II : accumulation ratio(Cmax) of Pregabalin | Pre-dose, 0,1,2,3,4,5,6,7,8,10,12,16,20,24,36 hours
Part II : accumulation ratio(AUCτ) of Pregabalin | Pre-dose, 0,1,2,3,4,5,6,7,8,10,12,16,20,24,36 hours

CONTACTS AND LOCATIONS:
Overall Officials: MinSoo Park, MD,PhD, Principal Investigator — Severance Hospital, Seoul, Korea
Locations (1):
- Severance Hospital, Seoul, Yonsei-ro Seodaemun-gu, South Korea